CLINICAL TRIAL: NCT00279565
Title: Randomized, Controlled Study of Buprenorphine and Methadone in Hepatitis C Patients in Need of Treatment
Brief Title: Buprenorphine Versus Methadone Maintenance in Hepatitis C Patients Receiving Peg-Intron and Rebetol (Study P04279)(TERMINATED)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial was terminated because of deviations from the protocol.
Sponsor: Indivior Inc. (Industry)
Collaborators: AESCA Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04279
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2007-02

CONDITIONS: Hepatitis C, Chronic
Keywords: buprenorphine; methadone; Peg-Intron; Rebetol
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Buprenorphine; Methadone; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: buprenorphine
Drug: methadone
Drug: pegylated interferon alfa-2b plus ribavirin

SUMMARY:
This randomized, single-center, controlled study is designed to evaluate the safety, tolerability, and efficacy of treatment with Peg-Intron with Rebetol in methadone or buprenorphine maintenance patients with hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with a history of intravenous drug abuse, who are willing to undergo methadone or buprenorphine substitution.
* Patients with newly diagnosed chronic hepatitis C.
* Age 18-65.
* Hepatitis C virus (HCV)-ribonucleic acid (RNA) positive in serum as measured by polymerase chain reaction (PCR) within the last 4 weeks.
* Genotype 2 or 3.
* Elevated alanine aminotransferase (ALT) levels.
* In women of child-bearing age, pregnancy must be excluded prior to entry into the study, and the use of a safe contraceptive device (intrauterine device, oral contraceptive, diaphragm + spermicide, condom + spermicide, tubal ligation) must be documented.
* Lab parameters:

  * Hemoglobin: >=12 g/dL (women) or >=13 g/dL (men)
  * Leukocytes >=3,000/µL
  * Thrombocytes >=100,000/µL
  * Prothrombin time (PT)/partial thromboplastin time (PTT)/coagulation within the normal range
  * Albumin: not more than 10% deviation from lower normal value
  * Thyroid-stimulating hormone (TSH) normal
  * Creatinine normal
  * Uric acid normal
  * Antinuclear antibodies <=1:160
* Signed informed consent.

Exclusion Criteria:

* Refusal by women of child-bearing age or by sexually active patients to use a safe contraceptive.
* Breast-feeding women.
* Cirrhosis stage B and C according to Child-Pugh.
* Signs of decompensated liver disease (ascites, bleeding varices and spontaneous encephalopathy).
* Confirmed co-infection with human immunodeficiency virus (HIV) or hepatitis B virus (HBV).
* Existing psychiatric comorbidity.
* Alcohol abuse.
* Active malignant disease or suspicion or history of malignant disease within five previous years (except for adequately treated basal cell carcinoma).
* Existing psoriasis or other dermatological disorder (relative exclusion criterion: due to great differences with regard to the severity of the disorder and the individual therapy compatibility, the therapy decision is at the discretion of the physician).
* Treatment with a study drug within the last 30 days.
* Any uncontrolled underlying medical conditions (e.g. diabetes).
* Clinically significant electrocardiogram (ECG) abnormalities and / or significant cardiovascular dysfunction within the last 6 months (angina, heart failure, recent myocardial infarction, severe hypertension or significant arrhythmia) is an exclusion criterion. In case of other suspected heart disease, a cardiologic examination is required prior to inclusion of the patient.
* Any liver disorder of other genesis than the study indication (with regard to elevated iron levels, only patients with manifest hemochromatosis are excluded).
* Autoimmune disorder (except LKM-positive patients: these patients may be included in the study).
* Misuse of buprenorphine or methadone.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128
Dates: Start 2005-08; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)